CLINICAL TRIAL: NCT04655833
Title: Integrative Korean Medicine Treatment for Inpatients With Failed Back Surgery Syndrome: A Retrospective Study With Survey
Status: Completed | Type: Observational
Sponsor: Jaseng Medical Foundation (Other)
Responsible Party: Principal Investigator, In-Hyuk Ha, KMD, Director, Jaseng Medical Foundation
Other Study IDs: JS-CT-2020-09-017
Record Dates: First submitted 2020-11-30; First posted 2020-12-07 (Actual); Last update posted 2021-01-20 (Actual); Status verified 2021-01

CONDITIONS: FBSS; Medicine, Korean Traditional
Keywords: acupuncture therapy; herbal medicine

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: phone survey — A questionnaire about the current symptoms and satisfaction for received treatment will be conducted over the phone for patients.

SUMMARY:
The purpose of this study is to reveal the effectiveness and safety of integrative Korean medicine for Failed Back Surgery Syndrome(FBSS) by observing inpatients treated with integrative Korean medicine.

This study is a retrospective observational study. The subjects for study are patients diagnosed with FBSS and who have been admitted to four Jaseng Hospital of Korean medicine (Gangnam, Bucheon, Daejeon, and Haeundae) for 2015.01.01-2019.12.31.

Medical records of selected patients will be analyzed, and telephone surveys will be conducted for each patient. The survey questions are Numeric ratinc scale (NRS), Oswestry Disability Index(ODI), quality of life, and Patient Global Impression of Change (PGIC), etc.

ELIGIBILITY:
Inclusion Criteria:

1. Patient who has a past history of lumbar surgery and has been hospitalized for persistent or recurrent pain and discomfort
2. Patient hospitalized for more than a week
3. Pateints above 19 years old and below 70 years old
4. Patients who have agreed to participate the study

Exclusion Criteria:

1. Patients who have been diagnosed with certain serious diseases that may cause back pain or limb pain (tumor metastases to the spine, spinal infections, ankylosing spondylitis(AS), acute fractures, spinal dislocation and so on)
2. Patients who have progressive neurological defects or severe synchronic neurological symptoms
3. The cause of the pain is soft tissue problems(tumor, fibromyalgia, rheumatoid arthritis, gout) and not related to spine
4. Patients who have been diagnosed with certain serious diseases that may cause disturbance to interpretation of conclusion (cardiovascular problems, kidney disease, diabetic neuropathy, dementia, epilepsy, and so on)
5. Patients who took steroids, immunosuppressants, psychiatric medications, or other drugs deemed inappropriate by researchers during hospitalization
6. Patient who has visited this medical institution within the last six months.
7. Patients deemed unable to participate in the clinical research by other researchers
8. Patients who haven't agreed to participate the study

Ages: 19 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The subjects for study are patients diagnosed with FBSS and who have been admitted to four Jaseng Hospital of Korean medicine (Gangnam, Bucheon, Daejeon, and Haeundae) for 2015.01.01-2019.12.31
Sampling Method: Non-Probability Sample
Enrollment: 106 (Actual)
Dates: Start 2020-10-22 (Actual); Primary Completion 2020-12-24 (Actual); Study Completion 2020-12-24 (Actual)

PRIMARY OUTCOMES:
Numeric rating scale (NRS) | Finish survey by November 2020
  NRS uses an 11-point scale to evaluate current neck pain and radiating pain where no pain is indicated by '0', and the worst pain imaginable by '10'. NRS was assessed at admission, 2 weeks after admission, discharge, and long term follow up.

SECONDARY OUTCOMES:
Oswestry Disability Index(ODI) | Finish survey by November 2020
  ODI is a 10-item questionnaire developed to evaluate the degree of disability for lower back pain. Each item is divided into 6 levels, and 0 to 5 points are awarded. The higher the score, the greater the degree of disability. We will conduct an validated Korean NDI questionnaire
The five level version of EuroQol-5 Dimension (EQ-5D) | Finish survey by November 2020
  EQ-5D is most widely used as a method of indirectly calculating the quality of life from various aspects. The EQ-5D-5L consists of 5 questions (mobility, self-care, usual activities, pain, anxiety/depression) that ask about the current state of health, and answers each question with 5 likert. (1=I have no problems about, 2=I have slight problems about, 3=I have moderate problems about, 4=I have severe problems about, 5=I am unable to about) In this study, the validated Korean version questionnaire will be used.
Patient Global Impression of Change (PGIC) | Finish survey by November 2020
  PGIC is an indicator that evaluates the improvement of patients in 7 steps, and the subject responds with improvement of functional limitation after treatment with 7 likert. (1=very much improved, 2=much improved, 3=minimally improved, 4=no change, 5=minimally worse, 6=much worse, 7=very much worse).
Spine surgery | Finish survey by November 2020
  The number of spinal surgery after discharge
Current symptoms survey | Finish survey by November 2020
  Pain, neurological problems, etc.
Treatment after discharge survey | Finish survey by November 2020
  Treatment history in the last 3 month
Satisfaction with integrative Korean medicine survey | Finish survey by November 2020
  Preference for integrative Korean medicine, satisfaction with integrative Korean medicine, How helpful hospitalization has been for returning to work and adjusting to daily life.

CONTACTS AND LOCATIONS:
Locations (1):
- Jaseng Medical Foundation, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No